CLINICAL TRIAL: NCT00985751
Title: Safety, Reactogenicity and Immunogenicity of GlaxoSmithKline (GSK) Biologicals' Investigational Vaccination Regimen in Children Aged 12-23 Months at the Time of First Vaccination.
Brief Title: Safety & Immunogenicity of Pneumococcal Vaccine 2189242A in Children Aged 12-23 Months at the Time of First Vaccination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 113171; 2009-012701-19 (EudraCT Number)
Record Dates: First submitted 2009-09-24; First posted 2009-09-28 (Estimated); Results first posted 2017-10-06 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Infections, Streptococcal
Keywords: immunogenicity; toddlers; Pneumococcal vaccine; Haemophilus influenzae; safety; Streptococcus pneumoniae; Streptococcus Pneumoniae Vaccines
MeSH Terms: conditions — Streptococcal Infections; Haemophilus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Group 1 (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK2189242A (formulation 1)
- Group 2 (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK2189242A (formulation 2)
- Group 3 (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK2189242A combined with pneumococcal vaccine GSK1024850A (formulation 3)
- Group 4 (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK2189242A combined with pneumococcal vaccine GSK1024850A (formulation 4)
- Control Group (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK1024850A

INTERVENTIONS:
Biological: Pneumococcal vaccine GSK2189242A (formulation 1) — Three doses will be administered intramuscularly, at Month 0, 2 and 6.
  Arms: Group 1
Biological: Pneumococcal vaccine GSK2189242A (formulation 2) — Three doses will be administered intramuscularly, at Month 0, 2 and 6
  Arms: Group 2
Biological: Pneumococcal vaccine GSK2189242A combined with pneumococcal vaccine GSK1024850A (formulation 3) — Three doses will be administered intramuscularly, at Month 0, 2 and 6
  Arms: Group 3
Biological: Pneumococcal vaccine GSK2189242A combined with pneumococcal vaccine GSK1024850A (formulation 4) — Three doses will be administered intramuscularly, at Month 0, 2 and 6
  Arms: Group 4
Biological: Pneumococcal vaccine GSK1024850A — Three doses will be administered intramuscularly, at Month 0, 2 and 6
  Arms: Control Group

SUMMARY:
This study will assess the safety, reactogenicity and immunogenicity of different formulations of GSK Biologicals' pneumococcal vaccine 2189242A when administered alone or in combination with the 10-valent pneumococcal conjugate vaccine (GSK1024850A vaccine) as a 2-dose primary vaccination course followed by a booster dose in healthy children aged 12-23 months at the time of first vaccination. Considering that febrile reactions are frequently observed following pneumococcal vaccination, usually co-administered with other routine paediatric vaccines, the primary study objective will focus on evaluating the increase in grade 3 fever (i.e. rectal temperature >40.0°C).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) (LAR) can and will comply with the requirements of the protocol
* Male or female between, and including, 12 and 23 months of age at the time of the first vaccination.
* Written informed consent obtained from the parents/LAR(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol during the study period starting from 30 days before each dose and ending 30 days after each dose of vaccine(s).
* Previous vaccination against S. pneumoniae since birth.
* History of any hypersensitivity reaction following any previous vaccination.
* Eczema and any history of allergy
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required), including human immunodeficiency virus infection.
* A family history of congenital or hereditary immunodeficiency.
* Major congenital defects or any chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease and/or fever at the time of enrolment.
* Fever is defined as temperature >= 37.5°C on oral or axillary setting, or >= 38.0°C on rectal setting.
* Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/ or any blood products within the 3 months preceding the first dose of study vaccine or planned use during the study period.
* Child in care.

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 257 (Actual)
Dates: Start 2009-11-24 (Actual); Primary Completion 2010-10-12 (Actual); Study Completion 2011-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- Czechia (9):
  - GSK Investigational Site, Chomutov
  - GSK Investigational Site, Děčín
  - GSK Investigational Site, Náchod
  - GSK Investigational Site, Odolena Voda
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Znojmo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=4501

REFERENCES:
- [Background] Prymula R, Pazdiora P, Traskine M, Ruggeberg JU, Borys D. Safety and immunogenicity of an investigational vaccine containing two common pneumococcal proteins in toddlers: a phase II randomized clinical trial. Vaccine. 2014 May 23;32(25):3025-34. doi: 10.1016/j.vaccine.2014.03.066. Epub 2014 Apr 1. PMID 24699466
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 113171 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113171 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113171 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113171 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113171 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- GSK 2189242A-LD Group: Subjects received 2 primary vaccination doses of GSK Biologicals' candidate pneumococcal protein vaccine (GSK 2189242A) containing the pneumococcal proteins dPly and PhtD, Low Dose (LD) vaccine formulation, at Month 0 and Month 2 and a booster dose at Month 6. The vaccine was administered intramuscularly, into the deltoid muscle or into the anterolateral thigh (if the deltoid muscle size was not adequate).
- GSK 2189242A-HD Group: Subjects received 2 primary vaccination doses of GSK Biologicals' candidate pneumococcal protein vaccine (GSK 2189242A) containing the pneumococcal proteins dPly and PhtD, High Dose (HD) vaccine formulation, at Month 0 and Month 2 and a booster dose at Month 6. The vaccine was administered intramuscularly, into the deltoid muscle or into the anterolateral thigh (if the deltoid muscle size was not adequate).
- Synflorix/GSK 2189242A-LD Group: Subjects received 2 primary vaccination doses of Synflorix™ vaccine combined with the pneumococcal protein vaccine (GSK 2189242A) containing the pneumococcal proteins dPly and PhtD, Low Dose (LD) vaccine formulation, at Month 0 and Month 2 and a booster dose at Month 6. The vaccine was administered intramuscularly, into the deltoid muscle or into the anterolateral thigh (if the deltoid muscle size was not adequate).
- Synflorix/GSK 2189242A-HD Group: Subjects received 2 primary vaccination doses of Synflorix™ vaccine combined with the pneumococcal protein vaccine (GSK 2189242A) containing the pneumococcal proteins dPly and PhtD, High Dose (HD) vaccine formulation, at Month 0 and Month 2 and a booster dose at Month 6. The vaccine was administered intramuscularly, into the deltoid muscle or into the anterolateral thigh (if the deltoid muscle size was not adequate).
- Synflorix Group: Subjects received 2 primary vaccination doses of Synflorix™ vaccine at Month 0 and Month 2 and a booster dose at Month 6. The vaccine was administered intramuscularly, into the deltoid muscle or into the anterolateral thigh (if the deltoid muscle size was not adequate).
Period: Overall Study
Arm/Group | GSK 2189242A-LD Group | GSK 2189242A-HD Group | Synflorix/GSK 2189242A-LD Group | Synflorix/GSK 2189242A-HD Group | Synflorix Group
Started | 51 | 52 | 52 | 51 | 51
Completed | 51 | 52 | 52 | 51 | 50
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK 2189242A-LD Group | GSK 2189242A-HD Group | Synflorix/GSK 2189242A-LD Group | Synflorix/GSK 2189242A-HD Group | Synflorix Group | Total
Number analyzed (Participants) | 51 | 52 | 52 | 51 | 51 | 257
Age, Continuous [Mean (Standard Deviation); unit: Months] | 17 (3.6) | 16.7 (3.81) | 17.1 (4.03) | 16.8 (3.96) | 16.3 (4.18) | 16.78 (3.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 23 | 29 | 28 | 127
  Male | 26 | 30 | 29 | 22 | 23 | 130
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White-Caucasian/European heritage | 51 | 52 | 51 | 51 | 49 | 254
  White-Arabic/North African heritage | 0 | 0 | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Fever > 40.0°C (Rectal Temperature)
Description: The number of subjects with rectal temperature higher (>) than 40.0 degrees Celsius (°C) is reported.
Time Frame: Within 7 days (Day 0-Day 6) following at least one dose of the primary vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Groups:
- Synflorix/GSK 2189242A Group: This group included subjects from Synflorix/GSK 2189242A-LD and Synflorix/GSK 2189242A-HD groups for whom pooled analysis was conducted.
Arm/Group | Synflorix Group | Synflorix/GSK 2189242A Group
Number analyzed (Participants) | 51 | 103
Participants | 0 | 1
Statistical Analysis 1: Comparison: Synflorix Group vs Synflorix/GSK 2189242A Group; Fever >40°C-non-inferiority: To compare the 2 formulations of GSK Biologicals' S. pneumoniae protein containing vaccine (GSK 2189242A) combined with Synflorix™ vaccine (pooled groups) versus Synflorix™ vaccine (Synflorix/GSK 2189242A Group minus Synflorix Group) with respect to the percentage of subjects reporting fever > 40.0°C (rectal temperature) within 7 days after at least 1 dose of primary vaccination; Test type: Non-Inferiority or Equivalence — The 95% CI for the difference between groups in the percentage of subjects with rectal temperature > 40.0°C within the 7-day follow-up period following primary vaccination was computed for the Synflorix/GSK 2189242A Group minus Synflorix Group. No statistically significant difference between groups in rectal temperature >40.0°C would be detected if the 95% CIs included 0 and non-inferiority would; Difference in percentage = 0.97, 95% CI 2-sided [-6.1 to 5.32]

2. Primary Outcome: Number of Subjects With Fever > 40.0°C (Rectal Temperature)
Description: The number of subjects with rectal temperature higher (>) than 40.0 degrees Celsius (°C) is reported.
Time Frame: Within 7 days (Day 0-Day 6) following at least one dose of the primary vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- GSK 2189242A Group: This group included subjects from GSK 2189242A-LD and GSK 2189242A-HD groups for whom pooled analysis was conducted.
Arm/Group | Synflorix Group | GSK 2189242A Group
Number analyzed (Participants) | 51 | 103
Participants | 0 | 1
Statistical Analysis 1: Comparison: Synflorix Group vs GSK 2189242A Group; Fever >40°C-non-inferiority: To compare the 2 formulations of GSK Biologicals' S. pneumoniae protein containing vaccine GSK 2189242A (pooled groups) versus Synflorix™ vaccine (GSK 2189242A Group minus Synflorix Group) with respect to the percentage of subjects reporting fever > 40.0°C (rectal temperature) within 7 days after at least 1 dose of primary vaccination; Test type: Non-Inferiority or Equivalence — The 95% CI for the difference between groups in the percentage of subjects with rectal temperature > 40.0°C within the 7-day follow-up period following primary vaccination was computed for the GSK 2189242A Group minus Synflorix Group. No statistically significant difference between groups in rectal temperature >40.0°C would be detected if the 95% CIs included 0 and non-inferiority would be express; Difference in percentage = 0.97, 95% CI 2-sided [-6.1 to 5.32]

3. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling. Grade 3 pain was defined as crying when limb was moved/spontaneously painful. Grade 3 swelling/redness was defined as swelling/redness larger than (>) 30 millimeters (mm). "Any" is defined as incidence of the specified symptom regardless of intensity.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose (Dose 1, Dose 2 and Booster dose)
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented and with the symptom sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 2189242A-LD Group | GSK 2189242A-HD Group | Synflorix/GSK 2189242A-LD Group | Synflorix/GSK 2189242A-HD Group | Synflorix Group
Number analyzed (Participants) | 51 | 52 | 52 | 51 | 51
Participants
  Any Pain Dose 1 | 18 | 15 | 31 | 23 | 26
  Grade 3 Pain Dose 1 | 0 | 0 | 1 | 2 | 4
  Any Redness Dose 1 | 17 | 20 | 32 | 28 | 25
  Grade 3 Redness Dose 1 | 1 | 0 | 5 | 4 | 2
  Any Swelling Dose 1 | 8 | 5 | 19 | 17 | 19
  Grade 3 Swelling Dose 1 | 0 | 0 | 2 | 2 | 1
  Any Pain Dose 2: number analyzed (Participants) | 51 | 52 | 52 | 51 | 50
  Any Pain Dose 2 | 15 | 22 | 24 | 27 | 27
  Grade 3 Pain Dose 2: number analyzed (Participants) | 51 | 52 | 52 | 51 | 50
  Grade 3 Pain Dose 2 | 0 | 0 | 2 | 2 | 3
  Any Redness Dose 2: number analyzed (Participants) | 51 | 52 | 52 | 51 | 50
  Any Redness Dose 2 | 21 | 25 | 23 | 22 | 24
  Grade 3 Redness Dose 2: number analyzed (Participants) | 51 | 52 | 52 | 51 | 50
  Grade 3 Redness Dose 2 | 1 | 1 | 4 | 1 | 3
  Any Swelling Dose 2: number analyzed (Participants) | 51 | 52 | 52 | 51 | 50
  Any Swelling Dose 2 | 11 | 9 | 18 | 11 | 16
  Grade 3 Swelling Dose 2: number analyzed (Participants) | 51 | 52 | 52 | 51 | 50
  Grade 3 Swelling Dose 2 | 0 | 0 | 5 | 1 | 2
  Any Pain Booster: number analyzed (Participants) | 51 | 51 | 52 | 51 | 50
  Any Pain Booster | 18 | 22 | 32 | 26 | 25
  Grade 3 Pain Booster: number analyzed (Participants) | 51 | 51 | 52 | 51 | 50
  Grade 3 Pain Booster | 0 | 0 | 3 | 2 | 1
  Any Redness Booster: number analyzed (Participants) | 51 | 51 | 52 | 51 | 50
  Any Redness Booster | 19 | 20 | 28 | 22 | 21
  Grade 3 Redness Booster: number analyzed (Participants) | 51 | 51 | 52 | 51 | 50
  Grade 3 Redness Booster | 2 | 2 | 5 | 4 | 3
  Any Swelling Booster: number analyzed (Participants) | 51 | 51 | 52 | 51 | 50
  Any Swelling Booster | 11 | 8 | 18 | 15 | 13
  Grade 3 Swelling Booster: number analyzed (Participants) | 51 | 51 | 52 | 51 | 50
  Grade 3 Swelling Booster | 0 | 3 | 3 | 1 | 3

4. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed include drowsiness, fever (defined as rectally temperature ≥ 38.0°C), irritability, and loss of appetite. Grade 3 drowsiness = drowsiness which prevented normal everyday activities. Grade 3 fever was defined as fever (rectally temperature) above (>) 40.0 degree Celsius (°C). Grade 3 irritability = crying that could not be comforted/preventing normal activity. Grade 3 loss of appetite = not eating at all. "Any" is defined as incidence of the specified symptom regardless of intensity or relationship to study vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose (Dose 1, Dose 2, Booster dose)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 2189242A-LD Group | GSK 2189242A-HD Group | Synflorix/GSK 2189242A-LD Group | Synflorix/GSK 2189242A-HD Group | Synflorix Group
Number analyzed (Participants) | 51 | 52 | 52 | 51 | 51
Participants
  Any Drowsiness Dose 1 | 16 | 13 | 24 | 20 | 26
  Grade 3 Drowsiness Dose 1 | 0 | 0 | 0 | 0 | 0
  Related Drowsiness Dose 1 | 6 | 6 | 13 | 10 | 16
  Any Irritability Dose 1 | 21 | 16 | 31 | 27 | 23
  Grade 3 Irritability Dose 1 | 0 | 0 | 0 | 0 | 0
  Related Irritability Dose 1 | 6 | 9 | 17 | 16 | 14
  Any Loss of appetite Dose 1 | 15 | 7 | 14 | 12 | 14
  Grade 3 Loss of appetite Dose 1 | 2 | 0 | 1 | 0 | 0
  Related Loss of appetite Dose 1 | 4 | 5 | 9 | 3 | 7
  Any Fever Dose 1 | 7 | 8 | 14 | 12 | 12
  Grade 3 Fever Dose 1 | 0 | 1 | 1 | 0 | 0
  Related Fever Dose 1 | 3 | 2 | 7 | 8 | 9
  Any Drowsiness Dose 2: number analyzed (Participants) | 51 | 52 | 52 | 51 | 50
  Any Drowsiness Dose 2 | 12 | 16 | 17 | 15 | 23
  Grade 3 Drowsiness Dose 2: number analyzed (Participants) | 51 | 52 | 52 | 51 | 50
  Grade 3 Drowsiness Dose 2 | 0 | 0 | 0 | 0 | 0
  Related Drowsiness Dose 2: number analyzed (Participants) | 51 | 52 | 52 | 51 | 50
  Related Drowsiness Dose 2 | 6 | 11 | 11 | 10 | 18
  Any Irritability Dose 2: number analyzed (Participants) | 51 | 52 | 52 | 51 | 50
  Any Irritability Dose 2 | 12 | 18 | 22 | 24 | 27
  Grade 3 Irritability Dose 2: number analyzed (Participants) | 51 | 52 | 52 | 51 | 50
  Grade 3 Irritability Dose 2 | 0 | 0 | 0 | 0 | 1
  Related Irritability Dose 2: number analyzed (Participants) | 51 | 52 | 52 | 51 | 50
  Related Irritability Dose 2 | 3 | 11 | 17 | 18 | 21
  Any Loss of appetite Dose 2: number analyzed (Participants) | 51 | 52 | 52 | 51 | 50
  Any Loss of appetite Dose 2 | 8 | 10 | 12 | 9 | 13
  Grade 3 Loss of appetite Dose 2: number analyzed (Participants) | 51 | 52 | 52 | 51 | 50
  Grade 3 Loss of appetite Dose 2 | 1 | 0 | 0 | 0 | 0
  Related Loss of appetite Dose 2: number analyzed (Participants) | 51 | 52 | 52 | 51 | 50
  Related Loss of appetite Dose 2 | 4 | 5 | 9 | 5 | 7
  Any Fever Dose 2: number analyzed (Participants) | 51 | 52 | 52 | 51 | 50
  Any Fever Dose 2 | 9 | 12 | 8 | 9 | 7
  Grade 3 Fever Dose 2: number analyzed (Participants) | 51 | 52 | 52 | 51 | 50
  Grade 3 Fever Dose 2 | 0 | 0 | 0 | 0 | 0
  Related Fever Dose 2: number analyzed (Participants) | 51 | 52 | 52 | 51 | 50
  Related Fever Dose 2 | 2 | 6 | 5 | 7 | 7
  Any Drowsiness Booster: number analyzed (Participants) | 51 | 51 | 52 | 51 | 50
  Any Drowsiness Booster | 13 | 13 | 18 | 12 | 17
  Grade 3 Drowsiness Booster: number analyzed (Participants) | 51 | 51 | 52 | 51 | 50
  Grade 3 Drowsiness Booster | 0 | 0 | 0 | 0 | 0
  Related Drowsiness Booster: number analyzed (Participants) | 51 | 51 | 52 | 51 | 50
  Related Drowsiness Booster | 7 | 9 | 11 | 10 | 11
  Any Irritability Booster: number analyzed (Participants) | 51 | 51 | 52 | 51 | 50
  Any Irritability Booster | 15 | 17 | 26 | 17 | 19
  Grade 3 Irritability Booster: number analyzed (Participants) | 51 | 51 | 52 | 51 | 50
  Grade 3 Irritability Booster | 0 | 0 | 0 | 1 | 1
  Related Irritability Booster: number analyzed (Participants) | 51 | 51 | 52 | 51 | 50
  Related Irritability Booster | 9 | 11 | 15 | 13 | 13
  Any Loss of appetite Booster: number analyzed (Participants) | 51 | 51 | 52 | 51 | 50
  Any Loss of appetite Booster | 6 | 10 | 13 | 15 | 8
  Grade 3 Loss of appetite Booster: number analyzed (Participants) | 51 | 51 | 52 | 51 | 50
  Grade 3 Loss of appetite Booster | 2 | 0 | 1 | 1 | 1
  Related Loss of appetite Booster: number analyzed (Participants) | 51 | 51 | 52 | 51 | 50
  Related Loss of appetite Booster | 4 | 4 | 7 | 7 | 6
  Any Fever Booster: number analyzed (Participants) | 51 | 51 | 52 | 51 | 50
  Any Fever Booster | 8 | 10 | 10 | 5 | 7
  Grade 3 Fever Booster: number analyzed (Participants) | 51 | 51 | 52 | 51 | 50
  Grade 3 Fever Booster | 0 | 0 | 0 | 0 | 0
  Related Fever Booster: number analyzed (Participants) | 51 | 51 | 52 | 51 | 50
  Related Fever Booster | 5 | 3 | 7 | 2 | 3

5. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. "Any" is defined an incidence of an unsolicited AE regardless of intensity or relationship to study vaccination.
Time Frame: During the 31-day (Days 0-30) follow-up period after each primary dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 2189242A-LD Group | GSK 2189242A-HD Group | Synflorix/GSK 2189242A-LD Group | Synflorix/GSK 2189242A-HD Group | Synflorix Group
Number analyzed (Participants) | 51 | 52 | 52 | 51 | 51
Participants | 25 | 24 | 31 | 24 | 22

6. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: as for outcome 5
Time Frame: During the 31-day (Days 0-30) follow-up period after the booster dose
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 2189242A-LD Group | GSK 2189242A-HD Group | Synflorix/GSK 2189242A-LD Group | Synflorix/GSK 2189242A-HD Group | Synflorix Group
Number analyzed (Participants) | 51 | 51 | 52 | 51 | 50
Participants | 14 | 12 | 13 | 4 | 9

7. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period starting at the administration of the first vaccine dose up to study end (from Day 0 up to Month 7)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 2189242A-LD Group | GSK 2189242A-HD Group | Synflorix/GSK 2189242A-LD Group | Synflorix/GSK 2189242A-HD Group | Synflorix Group
Number analyzed (Participants) | 51 | 52 | 52 | 51 | 51
Participants | 5 | 3 | 5 | 0 | 4

8. Secondary Outcome: Anti-pneumococcal dPly and PhtD Proteins Antibody Concentrations
Description: Seropositivity status, defined as anti-pneumococcal dPly antibody concentrations ≥ 599 Luminex Units per milliliter (LU/mL) and anti-pneumococcal PhtD antibody concentrations ≥ 391 LU/mL.
Time Frame: One month post-dose 2 (Month 3), prior to the booster dose (Month 6) and one month post-booster (Month 7)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available.
Measure: Geometric Mean (95% Confidence Interval); unit: LU/mL
Arm/Group | GSK 2189242A-LD Group | GSK 2189242A-HD Group | Synflorix/GSK 2189242A-LD Group | Synflorix/GSK 2189242A-HD Group | Synflorix Group
Number analyzed (Participants) | 45 | 45 | 47 | 41 | 41
LU/mL
  Anti-dPly, Post-dose 2: number analyzed (Participants) | 45 | 43 | 45 | 39 | 41
  Anti-dPly, Post-dose 2 | 135703.5 [95376.62 to 193081.3] | 148447.5 [101599.9 to 216896.7] | 32436.07 [25523.77 to 41220.35] | 57149.83 [44908.69 to 72727.64] | 3759.82 [2376.77 to 5947.68]
  Anti-dPly, Pre-booster: number analyzed (Participants) | 44 | 45 | 46 | 40 | 40
  Anti-dPly, Pre-booster | 100811.4 [74005.55 to 137326.8] | 96552.52 [73753.5 to 126399.3] | 19573.55 [14948.37 to 25629.82] | 29592.91 [22065.25 to 39688.66] | 4654.16 [2879.42 to 7522.78]
  Anti-dPly, Post-booster: number analyzed (Participants) | 44 | 43 | 47 | 41 | 41
  Anti-dPly, Post-booster | 224726.2 [178187.6 to 283419.8] | 305912.3 [248087.9 to 377214.4] | 44123.43 [34299.98 to 56760.29] | 85805.02 [67740.53 to 108686.8] | 4553.43 [2878.04 to 7204.12]
  Anti-PhtD, Post-dose 2: number analyzed (Participants) | 45 | 43 | 45 | 39 | 41
  Anti-PhtD, Post-dose 2 | 30402.84 [20723.61 to 44602.88] | 35043.91 [24164.16 to 50822.19] | 23438.06 [16617.86 to 33057.36] | 22141.18 [15065.44 to 32540.15] | 3795.68 [2268.23 to 6351.73]
  Anti-PhtD, Pre-booster: number analyzed (Participants) | 44 | 45 | 46 | 40 | 40
  Anti-PhtD, Pre-booster | 24350.58 [17056.09 to 34764.74] | 23918.77 [17724.59 to 32277.63] | 14375.59 [9338.31 to 22130.1] | 12721.01 [8498 to 19042.62] | 4814.97 [2881.25 to 8046.46]
  Anti-PhtD, Post-booster: number analyzed (Participants) | 44 | 43 | 47 | 41 | 41
  Anti-PhtD, Post-booster | 65584.24 [50985.27 to 84363.43] | 77312.07 [58589.49 to 102017.6] | 32609.19 [23615.58 to 45027.88] | 36098.18 [26620.97 to 48949.34] | 5072.43 [3023.97 to 8508.53]

9. Secondary Outcome: Anti-pneumococcal Serotypes and Cross-reactive Serotypes Antibody Concentrations
Description: Seropositivity status, defined as anti-pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F and cross-reactive serotype 6A and 19 antibody concentrations ≥ 0.05 microgram per milliliter (µg/mL).
Time Frame: One month post-dose 2 (Month 3), prior to the booster dose (Month 6) and one month post-booster (Month 7)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GSK 2189242A-LD Group | GSK 2189242A-HD Group | Synflorix/GSK 2189242A-LD Group | Synflorix/GSK 2189242A-HD Group | Synflorix Group
Number analyzed (Participants) | 43 | 44 | 47 | 41 | 41
µg/mL
  Anti-1, Post-Dose 2: number analyzed (Participants) | 40 | 36 | 46 | 40 | 41
  Anti-1, Post-Dose 2 | 0.04 [0.03 to 0.05] | 0.05 [0.04 to 0.06] | 2.5 [2.01 to 3.11] | 2.08 [1.56 to 2.77] | 2.13 [1.62 to 2.79]
  Anti-1, Pre-booster: number analyzed (Participants) | 43 | 42 | 45 | 40 | 40
  Anti-1, Pre-booster | 0.05 [0.03 to 0.06] | 0.05 [0.04 to 0.07] | 0.87 [0.68 to 1.12] | 0.75 [0.57 to 0.99] | 0.73 [0.55 to 0.97]
  Anti-1, Post-booster: number analyzed (Participants) | 40 | 41 | 47 | 41 | 41
  Anti-1, Post-booster | 0.04 [0.03 to 0.06] | 0.05 [0.04 to 0.08] | 2.69 [2.13 to 3.39] | 2.47 [2.03 to 3] | 2.4 [1.85 to 3.12]
  Anti-4, Post-Dose 2: number analyzed (Participants) | 37 | 37 | 46 | 40 | 41
  Anti-4, Post-Dose 2 | 0.05 [0.03 to 0.08] | 0.03 [0.02 to 0.03] | 6.42 [5.23 to 7.87] | 6.6 [5.12 to 8.52] | 5.67 [4.56 to 7.06]
  Anti-4, Pre-booster: number analyzed (Participants) | 41 | 41 | 46 | 41 | 40
  Anti-4, Pre-booster | 0.05 [0.03 to 0.07] | 0.03 [0.03 to 0.03] | 2.3 [1.82 to 2.91] | 2.36 [1.79 to 3.11] | 2.11 [1.68 to 2.64]
  Anti-4, Post-booster: number analyzed (Participants) | 40 | 41 | 47 | 41 | 41
  Anti-4, Post-booster | 0.05 [0.03 to 0.07] | 0.04 [0.03 to 0.05] | 5.26 [4.14 to 6.69] | 5.61 [4.46 to 7.07] | 5.18 [4.05 to 6.63]
  Anti-5, Post-Dose 2: number analyzed (Participants) | 31 | 34 | 44 | 39 | 41
  Anti-5, Post-Dose 2 | 0.06 [0.04 to 0.08] | 0.06 [0.05 to 0.08] | 2.42 [1.85 to 3.17] | 2.41 [1.85 to 3.13] | 2.36 [1.88 to 2.97]
  Anti-5, Pre-booster: number analyzed (Participants) | 42 | 43 | 45 | 41 | 40
  Anti-5, Pre-booster | 0.07 [0.05 to 0.1] | 0.06 [0.05 to 0.08] | 1.08 [0.83 to 1.41] | 1.05 [0.81 to 1.36] | 1.18 [0.94 to 1.48]
  Anti-5, Post-booster: number analyzed (Participants) | 41 | 43 | 47 | 41 | 41
  Anti-5, Post-booster | 0.07 [0.05 to 0.09] | 0.07 [0.05 to 0.09] | 3.57 [2.79 to 4.57] | 3.45 [2.7 to 4.41] | 3.84 [2.98 to 4.95]
  Anti-6B, Post-Dose 2: number analyzed (Participants) | 43 | 39 | 46 | 40 | 41
  Anti-6B, Post-Dose 2 | 0.04 [0.03 to 0.05] | 0.03 [0.02 to 0.03] | 0.55 [0.37 to 0.81] | 0.48 [0.32 to 0.72] | 0.55 [0.39 to 0.78]
  Anti-6B, Pre-booster: number analyzed (Participants) | 42 | 41 | 44 | 40 | 40
  Anti-6B, Pre-booster | 0.04 [0.03 to 0.05] | 0.04 [0.03 to 0.05] | 0.39 [0.28 to 0.54] | 0.42 [0.3 to 0.59] | 0.46 [0.34 to 0.62]
  Anti-6B, Post-booster: number analyzed (Participants) | 41 | 42 | 47 | 41 | 40
  Anti-6B, Post-booster | 0.04 [0.03 to 0.06] | 0.04 [0.03 to 0.06] | 1.08 [0.74 to 1.57] | 1.14 [0.83 to 1.57] | 1.08 [0.78 to 1.52]
  Anti-7F, Post-Dose 2: number analyzed (Participants) | 37 | 38 | 46 | 40 | 41
  Anti-7F, Post-Dose 2 | 0.04 [0.03 to 0.06] | 0.04 [0.03 to 0.04] | 5.03 [4.16 to 6.09] | 4.73 [3.89 to 5.74] | 3.72 [3.17 to 4.36]
  Anti-7F, Pre-booster: number analyzed (Participants) | 42 | 44 | 46 | 41 | 40
  Anti-7F, Pre-booster | 0.04 [0.03 to 0.06] | 0.03 [0.03 to 0.04] | 2.6 [2.14 to 3.15] | 2.36 [1.94 to 2.86] | 2.14 [1.82 to 2.51]
  Anti-7F, Post-booster: number analyzed (Participants) | 41 | 43 | 47 | 41 | 41
  Anti-7F, Post-booster | 0.04 [0.03 to 0.06] | 0.04 [0.03 to 0.05] | 5.9 [4.83 to 7.2] | 5.25 [4.36 to 6.32] | 4.65 [3.77 to 5.72]
  Anti-9V, Post-Dose 2: number analyzed (Participants) | 42 | 40 | 46 | 40 | 41
  Anti-9V, Post-Dose 2 | 0.04 [0.03 to 0.06] | 0.03 [0.02 to 0.03] | 2.81 [2.24 to 3.51] | 2.49 [1.95 to 3.19] | 1.55 [1.21 to 2]
  Anti-9V, Pre-booster: number analyzed (Participants) | 41 | 42 | 45 | 41 | 40
  Anti-9V, Pre-booster | 0.04 [0.03 to 0.05] | 0.03 [0.03 to 0.04] | 1.44 [1.15 to 1.81] | 1.26 [0.94 to 1.67] | 0.95 [0.73 to 1.24]
  Anti-9V, Post-booster: number analyzed (Participants) | 39 | 40 | 47 | 41 | 40
  Anti-9V, Post-booster | 0.04 [0.03 to 0.06] | 0.03 [0.02 to 0.04] | 3.13 [2.48 to 3.93] | 3.21 [2.45 to 4.19] | 2.18 [1.71 to 2.79]
  Anti-14, Post-Dose 2: number analyzed (Participants) | 43 | 36 | 46 | 40 | 41
  Anti-14, Post-Dose 2 | 0.1 [0.07 to 0.14] | 0.09 [0.06 to 0.14] | 5.18 [3.91 to 6.86] | 3.78 [2.92 to 4.91] | 4.63 [3.71 to 5.77]
  Anti-14, Pre-booster: number analyzed (Participants) | 40 | 40 | 46 | 40 | 40
  Anti-14, Pre-booster | 0.11 [0.08 to 0.17] | 0.11 [0.07 to 0.18] | 2.86 [2.25 to 3.65] | 2.3 [1.81 to 2.91] | 2.71 [2.17 to 3.38]
  Anti-14, Post-booster: number analyzed (Participants) | 42 | 43 | 47 | 41 | 41
  Anti-14, Post-booster | 0.13 [0.09 to 0.18] | 0.16 [0.1 to 0.26] | 7.74 [6.03 to 9.94] | 6.62 [5.22 to 8.4] | 5.98 [4.68 to 7.63]
  Anti-18C, Post-Dose 2: number analyzed (Participants) | 39 | 39 | 45 | 40 | 41
  Anti-18C, Post-Dose 2 | 0.04 [0.03 to 0.06] | 0.04 [0.03 to 0.05] | 13.92 [10.75 to 18.03] | 16.92 [13.61 to 21.03] | 12.56 [9.8 to 16.1]
  Anti-18C, Pre-booster: number analyzed (Participants) | 41 | 42 | 45 | 41 | 40
  Anti-18C, Pre-booster | 0.05 [0.03 to 0.07] | 0.04 [0.03 to 0.05] | 4.94 [3.83 to 6.38] | 5.51 [4.3 to 7.05] | 4.79 [3.69 to 6.21]
  Anti-18C, Post-booster: number analyzed (Participants) | 42 | 44 | 47 | 41 | 40
  Anti-18C, Post-booster | 0.05 [0.03 to 0.07] | 0.05 [0.03 to 0.07] | 16.12 [12.2 to 21.32] | 21.98 [16.67 to 28.99] | 14.62 [10.9 to 19.6]
  Anti-19F, Post-Dose 2: number analyzed (Participants) | 33 | 35 | 45 | 39 | 41
  Anti-19F, Post-Dose 2 | 0.05 [0.03 to 0.08] | 0.06 [0.03 to 0.12] | 8.6 [6.37 to 11.63] | 10.08 [7.21 to 14.09] | 8.87 [6.2 to 12.7]
  Anti-19F, Pre-booster: number analyzed (Participants) | 38 | 40 | 46 | 41 | 40
  Anti-19F, Pre-booster | 0.06 [0.04 to 0.1] | 0.05 [0.03 to 0.09] | 4.15 [2.94 to 5.85] | 4.72 [3.54 to 6.3] | 4.33 [3.06 to 6.12]
  Anti-19F, Post-booster: number analyzed (Participants) | 41 | 40 | 47 | 41 | 41
  Anti-19F, Post-booster | 0.06 [0.04 to 0.09] | 0.07 [0.04 to 0.13] | 10.46 [7.35 to 14.88] | 14.38 [10.53 to 19.63] | 11.32 [7.94 to 16.13]
  Anti-23F, Post-Dose 2: number analyzed (Participants) | 38 | 38 | 45 | 39 | 41
  Anti-23F, Post-Dose 2 | 0.03 [0.03 to 0.04] | 0.04 [0.03 to 0.05] | 1.19 [0.82 to 1.74] | 0.91 [0.62 to 1.33] | 0.73 [0.54 to 0.98]
  Anti-23F, Pre-booster: number analyzed (Participants) | 42 | 41 | 45 | 41 | 40
  Anti-23F, Pre-booster | 0.03 [0.03 to 0.04] | 0.04 [0.03 to 0.06] | 0.71 [0.5 to 0.99] | 0.62 [0.45 to 0.85] | 0.51 [0.39 to 0.67]
  Anti-23F, Post-booster: number analyzed (Participants) | 41 | 43 | 47 | 41 | 40
  Anti-23F, Post-booster | 0.03 [0.03 to 0.04] | 0.05 [0.03 to 0.06] | 1.92 [1.42 to 2.6] | 2.04 [1.56 to 2.65] | 1.47 [1.04 to 2.06]
  Anti-6A, Post-Dose 2: number analyzed (Participants) | 33 | 37 | 43 | 40 | 41
  Anti-6A, Post-Dose 2 | 0.04 [0.03 to 0.07] | 0.03 [0.03 to 0.04] | 0.32 [0.2 to 0.51] | 0.27 [0.16 to 0.45] | 0.31 [0.2 to 0.48]
  Anti-6A, Pre-booster: number analyzed (Participants) | 42 | 42 | 44 | 41 | 40
  Anti-6A, Pre-booster | 0.04 [0.03 to 0.06] | 0.04 [0.03 to 0.04] | 0.24 [0.17 to 0.34] | 0.24 [0.15 to 0.38] | 0.27 [0.18 to 0.4]
  Anti-6A, Post-booster: number analyzed (Participants) | 42 | 40 | 47 | 41 | 40
  Anti-6A, Post-booster | 0.04 [0.03 to 0.06] | 0.04 [0.03 to 0.06] | 0.53 [0.35 to 0.79] | 0.56 [0.36 to 0.87] | 0.58 [0.37 to 0.9]
  Anti-19A, Post-Dose 2: number analyzed (Participants) | 33 | 35 | 43 | 39 | 41
  Anti-19A, Post-Dose 2 | 0.07 [0.04 to 0.12] | 0.05 [0.03 to 0.06] | 1.08 [0.71 to 1.62] | 0.97 [0.63 to 1.48] | 0.93 [0.61 to 1.43]
  Anti-19A, Pre-booster: number analyzed (Participants) | 43 | 42 | 44 | 41 | 40
  Anti-19A, Pre-booster | 0.07 [0.04 to 0.1] | 0.05 [0.04 to 0.06] | 0.85 [0.61 to 1.17] | 0.68 [0.47 to 0.98] | 0.62 [0.42 to 0.93]
  Anti-19A, Post-booster: number analyzed (Participants) | 41 | 39 | 47 | 41 | 41
  Anti-19A, Post-booster | 0.07 [0.05 to 0.11] | 0.05 [0.04 to 0.07] | 2.76 [1.92 to 3.96] | 2.98 [2.08 to 4.26] | 2.06 [1.3 to 3.25]

10. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Serotypes and Cross-reactive Serotypes
Description: Seropositivity status, defined as Opsonophagocytic activity against pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F and cross-reactive serotypes 6A and 19A ≥ 8.
Time Frame: One month post-dose 2 (Month 3), prior to the booster dose (Month 6) and one month post-booster (Month 7)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK 2189242A-LD Group | GSK 2189242A-HD Group | Synflorix/GSK 2189242A-LD Group | Synflorix/GSK 2189242A-HD Group | Synflorix Group
Number analyzed (Participants) | 35 | 36 | 37 | 36 | 37
Titers
  OPSONO-1, Post-Dose 2: number analyzed (Participants) | 27 | 33 | 35 | 30 | 30
  OPSONO-1, Post-Dose 2 | 4 [4 to 4] | 5.4 [3.8 to 7.8] | 71.8 [40.9 to 126.1] | 48.2 [26.5 to 87.6] | 90 [52.9 to 153]
  OPSONO-1, Pre-booster: number analyzed (Participants) | 35 | 35 | 33 | 35 | 34
  OPSONO-1, Pre-booster | 4 [4 to 4] | 4.3 [3.7 to 5] | 23 [13.1 to 40.3] | 12.4 [7.6 to 20.3] | 19.3 [11.1 to 33.6]
  OPSONO-1, Post-booster: number analyzed (Participants) | 31 | 35 | 37 | 36 | 37
  OPSONO-1, Post-booster | 5.2 [4 to 6.9] | 8.1 [4.8 to 13.7] | 169.5 [96.1 to 298.8] | 200 [138.2 to 289.4] | 206.9 [123.1 to 347.5]
  OPSONO-4, Post-Dose 2: number analyzed (Participants) | 20 | 29 | 32 | 29 | 29
  OPSONO-4, Post-Dose 2 | 7 [3.1 to 15.6] | 8.9 [4.5 to 17.6] | 1260.2 [856.1 to 1855.2] | 1197.9 [784.1 to 1830.2] | 1220.4 [913.8 to 1629.9]
  OPSONO-4, Pre-booster: number analyzed (Participants) | 28 | 29 | 29 | 33 | 30
  OPSONO-4, Pre-booster | 12.6 [5.6 to 28.4] | 16.2 [7 to 37.2] | 247.9 [117.4 to 523.2] | 259.9 [120.6 to 560] | 478.9 [309.3 to 741.3]
  OPSONO-4, Post-booster: number analyzed (Participants) | 24 | 31 | 35 | 32 | 34
  OPSONO-4, Post-booster | 15.5 [6.1 to 39.5] | 17.8 [7.3 to 43.4] | 1206.2 [888.9 to 1636.8] | 1385 [974.5 to 1968.4] | 1476 [1076 to 2024.6]
  OPSONO-5, Post-Dose 2: number analyzed (Participants) | 27 | 33 | 33 | 30 | 31
  OPSONO-5, Post-Dose 2 | 4 [4 to 4] | 4.7 [3.4 to 6.5] | 43.8 [27.1 to 70.8] | 37.3 [21.7 to 64] | 42 [26.6 to 66.4]
  OPSONO-5, Pre-booster: number analyzed (Participants) | 34 | 35 | 34 | 33 | 34
  OPSONO-5, Pre-booster | 4.5 [3.5 to 5.8] | 4 [4 to 4] | 12.8 [8.2 to 19.9] | 14.8 [9.6 to 23] | 17 [10.9 to 26.4]
  OPSONO-5, Post-booster: number analyzed (Participants) | 30 | 36 | 37 | 34 | 36
  OPSONO-5, Post-booster | 4 [4 to 4] | 5.1 [3.8 to 6.7] | 99.3 [62.1 to 158.8] | 110.4 [73.1 to 166.8] | 160.7 [113 to 228.7]
  OPSONO-6B, Post-Dose 2: number analyzed (Participants) | 16 | 21 | 27 | 25 | 28
  OPSONO-6B, Post-Dose 2 | 15 [4.2 to 53.1] | 23.4 [6.1 to 90.3] | 361.9 [120 to 1091.7] | 527.5 [202.6 to 1372.9] | 915.3 [543.4 to 1541.8]
  OPSONO-6B, Pre-booster: number analyzed (Participants) | 23 | 27 | 30 | 30 | 30
  OPSONO-6B, Pre-booster | 56.7 [16.2 to 198.4] | 61.6 [19.2 to 197.3] | 213.8 [79 to 578.1] | 513.1 [243.9 to 1079.6] | 371.9 [172.5 to 801.8]
  OPSONO-6B, Post-booster: number analyzed (Participants) | 24 | 33 | 33 | 34 | 35
  OPSONO-6B, Post-booster | 26.1 [7.7 to 88.7] | 30.8 [11.2 to 84.7] | 804.6 [343.5 to 1884.9] | 982.7 [527.6 to 1830.4] | 1523.1 [875.8 to 2649]
  OPSONO-7F, Post-Dose 2: number analyzed (Participants) | 27 | 33 | 33 | 29 | 30
  OPSONO-7F, Post-Dose 2 | 734.6 [369.7 to 1459.6] | 807.4 [445 to 1465.2] | 5703.7 [4143.6 to 7851.2] | 4936.6 [3320.7 to 7338.7] | 6154.4 [4244.4 to 8923.7]
  OPSONO-7F, Pre-booster: number analyzed (Participants) | 33 | 30 | 32 | 34 | 33
  OPSONO-7F, Pre-booster | 670.4 [317.5 to 1415.6] | 462.3 [187.5 to 1139.8] | 2450.1 [1637.4 to 3666.2] | 2713.5 [1836.1 to 4010.1] | 3844.5 [2725.7 to 5422.4]
  OPSONO-7F, Post-booster: number analyzed (Participants) | 30 | 35 | 35 | 33 | 36
  OPSONO-7F, Post-booster | 936.8 [510 to 1720.7] | 785.5 [428 to 1441.6] | 4109.3 [3086.9 to 5470.3] | 5730.4 [4262 to 7704.7] | 7404.7 [5271.1 to 10401.8]
  OPSONO-9V, Post-Dose 2: number analyzed (Participants) | 22 | 29 | 34 | 29 | 30
  OPSONO-9V, Post-Dose 2 | 26.5 [8.2 to 85.9] | 50.1 [17.5 to 143.7] | 4455 [2803.3 to 7079.9] | 3542.8 [2271.5 to 5525.5] | 3947.2 [2612.7 to 5963.5]
  OPSONO-9V, Pre-booster: number analyzed (Participants) | 30 | 28 | 32 | 33 | 32
  OPSONO-9V, Pre-booster | 172.4 [68.9 to 431.4] | 172 [57.6 to 513.2] | 2126.1 [1140.2 to 3964.4] | 2622.4 [1786.7 to 3849] | 3450 [2357.5 to 5048.7]
  OPSONO-9V, Post-booster: number analyzed (Participants) | 26 | 32 | 37 | 34 | 36
  OPSONO-9V, Post-booster | 173.5 [59.1 to 509.8] | 137.6 [51.7 to 366] | 4643.1 [3418.3 to 6306.9] | 5802.4 [4453 to 7560.8] | 6016.6 [4617.2 to 7840]
  OPSONO-14, Post-Dose 2: number analyzed (Participants) | 18 | 23 | 33 | 29 | 31
  OPSONO-14, Post-Dose 2 | 21.1 [6.7 to 66.8] | 11.9 [4.7 to 30.4] | 3324.8 [2324.8 to 4754.8] | 2580.7 [1788.4 to 3724] | 2487.6 [1703.4 to 3632.7]
  OPSONO-14, Pre-booster: number analyzed (Participants) | 30 | 30 | 32 | 34 | 33
  OPSONO-14, Pre-booster | 21 [8.5 to 51.6] | 27.9 [10.4 to 75.1] | 1390.5 [615.7 to 3140.4] | 1725.8 [972.1 to 3064] | 1776.6 [1009.5 to 3126.5]
  OPSONO-14, Post-booster: number analyzed (Participants) | 27 | 33 | 34 | 36 | 37
  OPSONO-14, Post-booster | 32.3 [11.5 to 90.9] | 46.7 [17 to 127.8] | 2911.6 [1841.3 to 4604] | 3729.8 [2693.2 to 5165.4] | 3094 [2353.3 to 4068]
  OPSONO-18C, Post-Dose 2: number analyzed (Participants) | 24 | 29 | 33 | 28 | 27
  OPSONO-18C, Post-Dose 2 | 4 [4 to 4] | 7.4 [3.7 to 15.1] | 1398.3 [810.6 to 2412] | 2538.4 [1787.3 to 3605] | 1905.4 [1271.4 to 2855.6]
  OPSONO-18C, Pre-booster: number analyzed (Participants) | 33 | 33 | 31 | 34 | 34
  OPSONO-18C, Pre-booster | 5.4 [3.4 to 8.3] | 5 [3.7 to 6.8] | 420.1 [192.8 to 915.3] | 1041 [699.6 to 1548.9] | 766.4 [468.4 to 1253.8]
  OPSONO-18C, Post-booster: number analyzed (Participants) | 26 | 32 | 34 | 32 | 33
  OPSONO-18C, Post-booster | 6 [3.3 to 10.7] | 8 [4.4 to 14.6] | 1764.6 [1243.6 to 2503.8] | 2640.6 [2083.3 to 3346.8] | 2123.4 [1493 to 3020.1]
  OPSONO-19F, Pre-booster: number analyzed (Participants) | 31 | 34 | 30 | 34 | 34
  OPSONO-19F, Pre-booster | 5 [3.1 to 8.2] | 8 [4.3 to 14.7] | 794.3 [476.6 to 1324] | 420.7 [197.4 to 896.4] | 625.4 [266.5 to 1467.7]
  OPSONO-19F, Post-booster: number analyzed (Participants) | 30 | 36 | 36 | 34 | 34
  OPSONO-19F, Post-booster | 4.9 [3.5 to 6.8] | 4.4 [3.7 to 5.2] | 173.3 [86.1 to 349] | 210.1 [118.4 to 373] | 260.7 [138 to 492.5]
  OPSONO-19F, Post-Dose 2: number analyzed (Participants) | 17 | 28 | 32 | 28 | 27
  OPSONO-19F, Post-Dose 2 | 5.6 [3.4 to 9.1] | 7.3 [4.3 to 12.6] | 1248.5 [740.4 to 2105.3] | 1823.7 [1252.9 to 2654.5] | 1625.3 [931.7 to 2835.3]
  OPSONO-23F, Post-Dose 2: number analyzed (Participants) | 20 | 28 | 34 | 28 | 29
  OPSONO-23F, Post-Dose 2 | 17.9 [5.1 to 62.9] | 107.8 [28.1 to 412.8] | 1735.5 [833.6 to 3613.3] | 3621.8 [2431.4 to 5395.2] | 2502.5 [1610.5 to 3888.6]
  OPSONO-23F, Pre-booster: number analyzed (Participants) | 30 | 33 | 32 | 33 | 33
  OPSONO-23F, Pre-booster | 23.2 [7.6 to 70.3] | 136.3 [36.1 to 514.6] | 989.7 [419.2 to 2336.8] | 1635.9 [691.7 to 3868.8] | 897.4 [381.6 to 2110.4]
  OPSONO-23F, Post-booster: number analyzed (Participants) | 25 | 33 | 35 | 35 | 36
  OPSONO-23F, Post-booster | 68.6 [17.3 to 271.2] | 106.7 [28.5 to 399.4] | 3598.5 [2422.2 to 5345.9] | 6108 [4335.9 to 8604.5] | 5296.1 [3857.9 to 7270.4]
  OPSONO-6A, Post-Dose 2: number analyzed (Participants) | 19 | 26 | 31 | 21 | 27
  OPSONO-6A, Post-Dose 2 | 9.3 [3.5 to 24.7] | 5.7 [3.4 to 9.5] | 225.3 [83.3 to 608.8] | 186.2 [55.3 to 627.2] | 364.5 [158.7 to 837.1]
  OPSONO-6A, Pre-booster: number analyzed (Participants) | 27 | 30 | 31 | 33 | 32
  OPSONO-6A, Pre-booster | 18.4 [7.6 to 44.5] | 9.4 [4.5 to 19.5] | 58.9 [21.6 to 160.3] | 99.4 [39.9 to 247.8] | 221.7 [93.8 to 524]
  OPSONO-6A, Post-booster: number analyzed (Participants) | 22 | 32 | 34 | 31 | 32
  OPSONO-6A, Post-booster | 11.8 [4.7 to 29.5] | 17.3 [7.9 to 37.9] | 308 [141 to 672.9] | 348.2 [154.9 to 782.5] | 554.3 [248.3 to 1237.6]
  OPSONO-19A, Post-Dose 2: number analyzed (Participants) | 25 | 31 | 34 | 28 | 29
  OPSONO-19A, Post-Dose 2 | 5.8 [3.4 to 9.9] | 4.6 [3.7 to 5.6] | 246 [109.7 to 551.7] | 363.2 [202.1 to 652.8] | 349.9 [177.1 to 691.6]
  OPSONO-19A, Pre-booster: number analyzed (Participants) | 35 | 35 | 33 | 35 | 32
  OPSONO-19A, Pre-booster | 6 [4 to 9.1] | 4.5 [3.8 to 5.3] | 56.7 [25.2 to 127.9] | 76.4 [36.3 to 160.7] | 87.8 [40.6 to 189.7]
  OPSONO-19A, Post-booster: number analyzed (Participants) | 30 | 36 | 34 | 34 | 34
  OPSONO-19A, Post-booster | 6.7 [4.3 to 10.3] | 6.3 [4.4 to 9.1] | 746.3 [407.8 to 1365.6] | 989.3 [652.5 to 1500] | 725.9 [367.8 to 1432.6]

11. Secondary Outcome: Antibody Concentrations to Protein D (Anti-PD)
Description: Seropositivity status, defined as anti-PD antibody concentrations ≥ 112 Luminex Units per milliliter (LU/mL).
Time Frame: One month post-dose 2 (Month 3), prior to the booster dose (Month 6) and one month post-booster (Month 7)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: LU/mL
Arm/Group | GSK 2189242A-LD Group | GSK 2189242A-HD Group | Synflorix/GSK 2189242A-LD Group | Synflorix/GSK 2189242A-HD Group | Synflorix Group
Number analyzed (Participants) | 45 | 45 | 47 | 41 | 41
LU/mL
  Anti-PD, Post-Dose 2: number analyzed (Participants) | 45 | 43 | 45 | 39 | 41
  Anti-PD, Post-Dose 2 | 90.9 [71.1 to 116.3] | 100.4 [76.3 to 132.1] | 1105.4 [833.7 to 1465.7] | 600.2 [426.5 to 844.7] | 860 [659.2 to 1121.9]
  Anti-PD, Pre-booster: number analyzed (Participants) | 44 | 45 | 46 | 40 | 40
  Anti-PD, Pre-booster | 89.1 [71.8 to 110.7] | 118.2 [89.6 to 155.9] | 734.6 [523.9 to 1030.1] | 463 [330.2 to 649.3] | 691.8 [527.6 to 907.1]
  Anti-PD, Post-booster: number analyzed (Participants) | 44 | 43 | 47 | 41 | 41
  Anti-PD, Post-booster | 97.9 [78 to 122.9] | 130.6 [93.1 to 183.3] | 1882.6 [1407.4 to 2518.1] | 1474.6 [1103.7 to 1970.3] | 1963.8 [1560.1 to 2472]

12. Secondary Outcome: Level of Anti-dPly Antibodies Inhibiting Ply Haemolysis Activity
Description: Inhibition of haemolysis activity of pneumolysin (Ply) by anti-dPly antibodies was measured in vitro by mean of a haemolytic assay. The haemolysis activity could be followed by measuring the level of haemoglobin released. Anti-dPly titers (for inhibition of haemolytic activity) ≥ 140.
Time Frame: One month post-dose 2 (Month 3), prior to the booster dose (Month 6) and one month post-booster (Month 7)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK 2189242A-LD Group | GSK 2189242A-HD Group | Synflorix/GSK 2189242A-LD Group | Synflorix/GSK 2189242A-HD Group | Synflorix Group
Number analyzed (Participants) | 43 | 38 | 43 | 39 | 40
Titers
  Anti-Hem-dPly, Post-Dose 2 | 3080 [2555.3 to 3712.5] | 2988.7 [2410.1 to 3706.2] | 1278.9 [1048.2 to 1560.3] | 1814 [1495.3 to 2200.8] | 913.2 [699.1 to 1192.8]
  Anti-Hem-dPly, Pre-booster: number analyzed (Participants) | 37 | 37 | 37 | 34 | 35
  Anti-Hem-dPly, Pre-booster | 2441.1 [1867.1 to 3191.7] | 2193.7 [1737.3 to 2770] | 1141.5 [950.6 to 1370.6] | 1344.2 [1087.6 to 1661.3] | 995.9 [788.3 to 1258.2]
  Anti-Hem-dPly, Post-booster: number analyzed (Participants) | 31 | 32 | 36 | 32 | 30
  Anti-Hem-dPly, Post-booster | 4332.4 [3327.6 to 5640.4] | 5931.9 [4744.5 to 7416.4] | 1346.2 [1068.2 to 1696.5] | 2388.3 [1830.6 to 3115.9] | 818.6 [662.5 to 1011.5]

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-primary and post-booster vaccination period; Unsolicited AEs: during the 31-day (Days 0-30) post-primary and post-booster vaccination period; SAEs: during the whole study period (from Day 0 up to Month 7).
Arm/Group | GSK 2189242A-LD Group | GSK 2189242A-HD Group | Synflorix/GSK 2189242A-LD Group | Synflorix/GSK 2189242A-HD Group | Synflorix Group
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/52 | 0/52 | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 5/51 | 3/52 | 5/52 | 0/51 | 4/51
Other Adverse Events (participants affected / at risk) | 47/51 | 49/52 | 49/52 | 49/51 | 49/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK 2189242A-LD Group (N=51) | GSK 2189242A-HD Group (N=52) | Synflorix/GSK 2189242A-LD Group (N=52) | Synflorix/GSK 2189242A-HD Group (N=51) | Synflorix Group (N=51)
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Accidental exposure (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Open wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Affective disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pharyngo-tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK 2189242A-LD Group (N=51) | GSK 2189242A-HD Group (N=52) | Synflorix/GSK 2189242A-LD Group (N=52) | Synflorix/GSK 2189242A-HD Group (N=51) | Synflorix Group (N=51)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 2 | 1 | 4
Conjunctivitis (Eye disorders) | 0 | 0 | 3 | 0 | 0
Pain Primary (General disorders) | 27 | 28 | 34 | 33 | 34
Redness Primary (General disorders) | 24 | 30 | 36 | 33 | 30
Swelling Primary (General disorders) | 17 | 11 | 25 | 21 | 26
Pain Booster (General disorders) | 18 | 22 | 32 | 26 | 25
Redness Booster (General disorders) | 19 | 20 | 28 | 22 | 21
Swelling Booster (General disorders) | 11 | 8 | 18 | 15 | 13
Drowsiness Primary (General disorders) | 25 | 21 | 34 | 28 | 35
Irritability Primary (General disorders) | 26 | 23 | 35 | 36 | 35
Loss of appetite Primary (General disorders) | 19 | 15 | 20 | 19 | 23
Temperature/Rectally Primary (General disorders) | 13 | 16 | 18 | 18 | 17
Drowsiness Booster (General disorders) | 13 | 13 | 18 | 12 | 17
Irritability Booster (General disorders) | 15 | 17 | 26 | 17 | 19
Loss of appetite Booster (General disorders) | 6 | 10 | 13 | 15 | 8
Temperature/Rectally Booster (General disorders) | 8 | 10 | 10 | 5 | 7
Nasopharyngitis Primary (Infections and infestations) | 4 | 8 | 9 | 4 | 7
Nasopharyngitis Booster (Infections and infestations) | 3 | 3 | 2 | 0 | 2
Rhinitis Primary (Infections and infestations) | 3 | 1 | 4 | 1 | 1
Rhinitis Booster (Infections and infestations) | 4 | 1 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 3 | 4 | 4 | 3
Gastroenteritis (Infections and infestations) | 2 | 2 | 3 | 0 | 1
Viral infection (Infections and infestations) | 1 | 1 | 4 | 3 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 1 | 4 | 2
Varicella (Infections and infestations) | 0 | 1 | 1 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.